CLINICAL TRIAL: NCT01195961
Title: Facilitating Numerical Processing With Transcranial DC Stimulation in Developmental Dyscalculia
Brief Title: Facilitating Numerical Processing With Transcranial Stimulation in Developmental Dyscalculia
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100194; 10-N-0194
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-07-01

CONDITIONS: Cognition Disorder; Brain Mapping
Keywords: Direct Current Stimulation; Learning; Cognitive Enhancement; Cognitive Tasks; Cognitive Training; Developmental Dyscalculia; Learning Disability; Cognition Disorder
MeSH Terms: conditions — Cognition Disorders; Dyscalculia; Learning Disabilities

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Developmental dyscalculia is a learning disability in which individuals have difficulty learning or comprehending mathematics or other number concepts (such as keeping score during games, measuring time, or estimating distance). Developmental dyscalculia affects certain parts of the brain that are required for processing numbers. Research has shown that a form of brain stimulation called transcranial direct current stimulation (tDCS), applied when healthy individuals are being trained to carry out tasks with numbers, improved the ability to process numbers and solve math problems. More research is needed about whether tDCS can improve number processing in people with developmental dyscalculia.

Objectives:

- To examine whether the effects of transcranial direct current stimulation can help individuals with developmental dyscalculia perform mathematical calculations.

Eligibility:

- Individuals between 18 and 50 years of age who have been diagnosed with developmental dyscalculia, or are healthy volunteers without dyscalculia.

Design:

* Participants will have a screening visit and seven study visits. The screening visit and six of the study visits will take place consecutively over the course of 6 days, and the final visit will take place 3 months after the initial participation.
* Participants will be screened with a medical history, physical and neurological examination, and a brief examination to test for dyscalculia and determine the participant's dominant hand.
* Participants will be randomly assigned to one of two groups for the study. One group will receive tDCS during training to perform a task with numbers, and the other group will receive the same training with sham stimulation. Participants will not know which group they are in.
* During the study visits, participants will be trained on number tasks on 6 consecutive days. Before the tDCS or sham stimulation is applied at the beginning of the experiment and at the end of each training day, participants will perform other tasks with numbers. Participants will be evaluated based on the accuracy and speed with which they respond to the questions.
* At the followup visit, participants will perform the same number tasks they completed during the study visits. No tDCS will be performed at this visit.

DETAILED DESCRIPTION:
Objectives

Developmental dyscalculia (DD) is a condition in which subjects cannot process adequately numerical concepts. Performance of arithmetical calculations is associated with fMRI activity in an extended brain network that includes parietal and prefrontal cortices. Areas within the parietal lobe, required for numerical processing in healthy subjects, are abnormal in subjects with DD. The purpose of this single-blinded study is to determine if facilitatory transcranial direct current stimulation (tDCS) of these parietal areas in association with numerical training will improve processing of numerical information relative to sham in subjects with DD and in healthy volunteers.

Study population

30 healthy volunteers and 30 subjects with developmental dyscalculia (DD).

Design

Healthy volunteers and subjects with DD will be randomly assigned to one of two groups. Each group will receive anodal tDCS or sham with numerical training. All subjects will participate in 7 sessions. First, they will be trained on an ordinal numerical task (numerical training task) in which they will learn the magnitude relations between two numbers on 6 consecutive days while receiving sham stimulation or tDCS during the training. Subjects will see two numbers on the screen, one viewed on the left side of the screen and the other on the right side of the screen (example, 2, 4), and they have to decide which one is larger. Performance will be evaluated by fitting a power-law function. Before the beginning of the experiment and after each training day subjects will perform a numerical Stroop task that assesses the automaticity of numerical processing, and a number-space task that will provide information on the subject's accuracy of mapping numbers into space. At the end of each of the 6 training days (immediately post training) and 3 months (seventh session) later (retention measure) subjects will be tested on a dyscalculia test (The Dyscalculia Screener),the numerical Stroop task, and the number-space task

Outcome Measures

The primary outcome measure will be the improvement in automatic numerical processing (numerical Stroop task) as reflected by reaction times. Secondary outcomes are accuracy when mapping numbers into space (number-space task) and improvement in the dyscalculia score (Dyscalculia Screener).

ELIGIBILITY:
* INCLUSION CRITERIA:

We will include healthy volunteers and DD subjects who meet the following criteria:

Age 18 to 50 years

Able to provide informed consent

No history of math difficulties as determined by Dyscalculia Screener examination > upper 50th percentile (healthy volunteers)

Diagnosed with DD and scored < lower 25th percentile on Dyscalculia screening test (Developmental Dyscalculia subjects)

Edinburgh handedness inventory shows a laterality index (LI) > 75 (dexterity) or LI of less than -75 (left-handedness)

EXCLUSION CRITERIA:

We will exclude healthy volunteers and DD subjects if one of the following conditions applies:

Unable to perform the tasks due to visual problems

History of seizures or brain tumor

History of alcohol or drug abuse (defined as the use of a drug for a nontherapeutic effect ) or psychiatric illness such as severe depression

History of brain surgery

Drug treatment acting primarily on the central nervous system, which lowers the seizure threshold such as antipsychotic drugs (chlorprozamine, clozapine).

Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08-17; Study Completion 2011-07-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rubinsten O, Henik A. Developmental dyscalculia: heterogeneity might not mean different mechanisms. Trends Cogn Sci. 2009 Feb;13(2):92-9. doi: 10.1016/j.tics.2008.11.002. Epub 2009 Jan 8. PMID 19138550
- [Background] Cohen Kadosh R, Walsh V. Dyscalculia. Curr Biol. 2007 Nov 20;17(22):R946-7. doi: 10.1016/j.cub.2007.08.038. No abstract available. PMID 18029243
- [Background] von Aster MG, Shalev RS. Number development and developmental dyscalculia. Dev Med Child Neurol. 2007 Nov;49(11):868-73. doi: 10.1111/j.1469-8749.2007.00868.x. PMID 17979867